CLINICAL TRIAL: NCT06582628
Title: A Multicenter, Open Label, Randomized Phase II Trial to Evaluate the Efficacy of Talazoparib Plus Enzalutamide as First Line Treatment for Patients With Metastatic Castration Resistant Prostate Cancer Following Progression on Abiraterone
Brief Title: Talazoparib Plus Enzalutamide After Progression to Abiraterone in Metastatic Prostate Cancer: (TEAM PC)
Acronym: TEAM PC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Oncosur (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEAM PC_FOS06/2023; 2023-510536-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostatic Diseases; Prostatic Cancer; metastatic castration resistant prostate cancer (mCRPC); prostate adenocarcinoma; metastatic hormone-sensitive prostate cancer; Poly (ADP-ribose) Polymerases (PARP); Prostate Specific Antigen; Abiraterone
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases | interventions — enzalutamide; talazoparib

STUDY DESIGN:
Intervention Model Description: Exceptionally the Cross-over model will be allowed: from the control arm to the experimental arm upon progression is allowed in participants who meet certain criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Enzalutamide 160 mg orally daily continuously in 28-day cycles.
  Interventions: Drug: Enzalutamide capsule
- Enzalutamide and Talazoparib (Experimental): Enzalutamide 160 mg and Talazoparib 0.5 mg both orally daily and continuously in 28-day cycles.
  Interventions: Drug: Enzalutamide capsule and Talazoparib capsule

INTERVENTIONS:
Drug: Enzalutamide capsule — Enzalutamide capsules 160 mg orally daily
  Arms: Control
Drug: Enzalutamide capsule and Talazoparib capsule — Enzalutamide capsules 160 mg plus talazoparib capsules 0.5 mg, both orally daily
  Arms: Enzalutamide and Talazoparib

SUMMARY:
The purpose of this clinical trial is to determine the anti-tumor activity of talazoparib plus enzalutamide as first line treatment for metastatic castration resistant prostate cancer (mCRPC) in participants whose disease has progressed on abiraterone.

The main questions it aims to answer are:

* Does talazoparib plus enzalutamide improve efficacy in metastatic castration resistant prostate cancer (mCRPC) compared to enzalutamide alone?
* What is the time to disease progression [radiographic, Prostate Specific Antigen (PSA), clinical] in participants treated with talazoparib plus enzalutamide after progression on abiraterone?
* What medical problems do participants have when receiving talazoparib plus enzalutamide?

Researchers will compare the combination of talazoparib and enzalutamide as a first-line treatment for mCRPC to see if the combination improves the PSA response rate and delays progression compared to enzalutamide alone. The safety and tolerability of the combination (talazoparib and enzalutamide) will also be studied

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, phase II trial to evaluate the efficacy of the combination of talazoparib plus enzalutamide versus enzalutamide as first line treatment for metastatic castration resistant prostate cancer (mCRPC) in participants whose disease has progressed to abiraterone based treatment for metastatic hormone sensitive prostate cancer (mHSPC). Participants who meet the eligibility criteria will be randomized 1:1 to the experimental arm (enzalutamide and talazoparib) or control arm (enzalutamide) and will receive treatment until disease progression, unacceptable toxicity, death or discontinuation from the study treatment for any other reason.

Prostate cancer is the second most common malignancy in men worldwide with an estimated annual global incidence of 1.3 million and over 375,000 deaths. Aggressive variant prostate cancer is a clinically defined subset of metastatic castration resistant prostate cancers (mCRPC) characterized by the absence of response to androgen receptor (AR) targeted agents and neuroendocrine features. The treatments that are currently available are not effective, representing an unmet clinical need. The combination of talazoparib, a potent selective PARP inhibitor (PARPi) and enzalutamide (androgen receptor signaling inhibitor; ARSi) demonstrated in the TALAPRO-2 study improved efficacy in metastatic castration resistant prostate cancer (mCRPC) participants with and without DNA damage response (DDR) gene alterations as first line treatment (1L) compared to enzalutamide alone.

Up to 78 participants will be enrolled and randomized 1:1 to the experimental and control arms.Up to 19 participants will be allocated into the experimental arm in Stage 1. An interim analysis will be triggered once each patient on the experimental arm has been followed up for at least 16 weeks (or earlier if response status can be ascertained definitively) to decide whether to proceed to Stage 2 or discontinue the study. If greater than or equal to 6 responses are observed, recruitment will continue to Stage 2, enrolling 20 more participants on each arm; otherwise, the trial will stop.

Estimated duration of the study: 36 months. Accrual is expected to be completed in 18 months. Median treatment duration has been estimated in 10 months. After completion of (or discontinuation from) treatment, participants will be followed up for survival until end of study (EoS) that will occur at 18 months after the enrollment of the last patient included in the trial, unless premature termination of the study.

It is hypothesized that after progression to abiraterone, the addition of talazoparib to enzalutamide as 1L for mCRPC will result in improved PSA response rate and delayed progression compared to enzalutamide alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male age 18 or older.
2. Histological diagnosis of prostate adenocarcinoma without neuroendocrine differentiation or small cell features.
3. Willing and able to provide written informed consent to participate in the study. Written consent must be given before registration, according to International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) / Good clinical practice (GCP), and national/local regulations.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
5. Willing to provide tumor biopsies during the study. Note: At study entry, the pre-treatment fresh tumor biopsy could be replaced by an archived tumor biopsy upon agreement from the study chief investigator if such biopsy has been taken after progression to metastatic castration resistance and has both archived fresh-frozen material and a Formalin-fixed and paraffin-embedded (FFPE) block with a minimum tumor content more less than30 percent. Still the patient must be amenable and willing to undergo a new mandatory post-treatment biopsy.
6. Willing to provide blood samples for biomarker analysis.
7. Willing to give consent to sequencing of DNA damage repair (DDR) genes for analysis of the prevalence of somatic and germline aberrations in DNA damage repair genes.
8. Metastatic (M1) prostate cancer documented by bone scan, or soft tissue disease documented by computed tomography (CT), or magnetic resonance imaging (MRI).
9. Asymptomatic or minimally symptomatic prostate cancer at screening.
10. Estimated life expectancy of greater than or equal to 6 months from screening.
11. Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone (GnRH) agonist or antagonist for participants who have not undergone bilateral orchiectomy must be in place before screening and must continue throughout the study.

12 .Disease progression after at least 12 weeks of treatment with abiraterone for metastatic hormone-sensitive prostate cancer. Progression is defined as:

a. PSA rise of greater than or equal to 25 percent and an absolute increase of greater than or equal to 2 ng/mL above nadir (or baseline for participants with no PSA decline), confirmed by a second PSA value at least 3 weeks later.

and / or b. Limited radiographic progression: maximum of 2 new bone metastases, no new soft tissue metastasis and less than50percentincrease in the size of measurable soft tissue lesions.

13. Participants who have received prior docetaxel must meet the following criteria:

a. Received a maximum of 6 cycles of docetaxel for mHSPC. b. Received the last dose of docetaxel higher than 6 months prior to randomization.

14. Adequate organ function within 28 days before the first study treatment on Day 1, defined by the following:

1. Haemoglobin greater than or equal to 10 g/dL, no blood transfusions within 14 days before obtaining the haematology laboratory tests at screening,
2. Platelets greater than or equal to 100,000/μL no platelets transfusions within 14 days before obtaining the haematology laboratory tests at screening,
3. Neutrophils greater than or equal to 1500/μL, no growth factors given within 14 days before obtaining the haematology laboratory tests at screening,
4. Serum creatinine less than1.5X ULN or calculated creatinine clearance greater than or equal to 50 mL/min
5. Albumin greater than 3 g/dL,
6. AST or ALT less than 2.5 × ULN (less than 5 × ULN if liver function abnormalities are due to hepatic metastasis).
7. Total serum bilirubin less than 1.5 × ULN (less than 3 × ULN for participants with documented Gilbert syndrome or for whom indirect bilirubin concentrations suggest an extrahepatic source of elevation).

   15. Ability to swallow study medication tablets and comply with study requirements.

   16. Agrees to use a condom and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant, starting contraception at screening and continue throughout the study period and for 3 months after the final treatment administration, unless the patient is unable to maintain intercourse due to the androgen deprivation.

   17. Subjects must not donate sperm starting at screening and throughout the study period and for 3 months after the final abiraterone acetate administration.

   18. Subject agrees not to participate in another interventional study while on treatment.

   19. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Prior abiraterone treatment for less than 12 weeks or disease progression (either PSA or radiographic progression) within 6 months of starting abiraterone.
2. Disease progression less than 6 months after the last administration of docetaxel for mHSPC.
3. Known or suspected brain metastasis or active leptomeningeal disease.
4. A finding of superscan in a bone scan at screening. Superscan is defined as a bone scan which demonstrates markedly increased skeletal radioisotope uptake relative to soft tissues in association with absent or faint renal activity (absent kidney sign).
5. Symptomatic or impending spinal cord compression or cauda equina syndrome.
6. Use of opiate analgesia for pain from prostate cancer with average Brief pain inventory (BPI) questionnaire score higher than 6 and/or uncontrolled prostate cancer-related pain requiring increasing doses of opiates within 4 weeks prior to randomization
7. Prior treatment with an AR-targeted therapy (enzalutamide, apalutamide, darolutamide, ketoconazole) other than abiraterone for mHSPC; chemotherapy other than 6 cycles of docetaxel for mHSPC, immunotherapy or radiopharmaceuticals.
8. Therapeutic radiation therapy within, 14 days (7 days for limited-field palliative radiotherapy) prior to study enrolment, or participants who have not recovered from radiotherapy-related toxicities to grade less than or equal to 1 according to NCI-CTCAE v.5.0.
9. Major surgery within 4 weeks prior to randomization or participants who have not recovered from the side effects of any major surgery.
10. Administration of an investigational therapeutic or invasive surgical procedure (not including surgical castration) within 30 days of Cycle 1 Day 1 or currently enrolled in an investigational study.
11. History of seizure or any condition that may predispose to seizure (i.e., prior significant brain trauma, brain vascular malformation, etc) or subjects that have had an unexplained loss of consciousness or transient ischemic attacks within 1 year previous to scheduled day 1 of treatment.
12. Congenital long QT syndrome or ECG at screening with QT interval corrected using Fridericia's formula (QTcF) greater than 500 milliseconds.
13. articipants with clinically significant cardiovascular disease including but not limited to any of the following:

    1. Stroke, transient ischemic attack, unstable angina pectoris or documented myocardial infarction within 12 months prior to study entry.
    2. Symptomatic pericarditis or clinically significant pericardial effusion or myocarditis
    3. Documented congestive heart failure (New York Heart Association Class, NYHA functional classification III-IV)
    4. Uncontrolled, persistent hypertension defined as systolic blood pressure less than 170mmHg or diastolic blood pressure less than100mmHg. Subjects with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
14. Participants with any of the following cardiac conduction abnormalities: Ventricular arrhythmias except for benign premature ventricular contractions

    1. Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication.
    2. Conduction abnormality requiring a pacemaker.
    3. Other cardiac arrhythmia not controlled with medication.
15. Any clinically significant gastrointestinal disorder affecting absorption (i.e., extensive small bowel resection, active inflammatory bowel disease).
16. Active or symptomatic viral hepatitis or chronic liver disease.
17. Known/possible hypersensitivity, allergies to enzalutamide, talazoparib or any of capsule excipients.
18. Other malignancy except:

    1. Carcinoma in situ or non-melanoma skin cancer.
    2. A cancer diagnosed and treated greater than or equal to 5 years before randomization with no subsequent evidence of recurrence.
19. Any condition or situation which, in the opinion of the investigator, would put the subject at risk, may confound study results, or interfere with the subject's participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
PSA response (PSA50) | within the first 16 weeks
  Percentage of participants with a PSA decline greater than or equal to 50 percent from baseline confirmed by a consecutive PSA value (taken at least 3 weeks apart), prior to PSA progression
Objective response rate (ORR) | during the first 16 weeks
  Defined as the best overall radiographic response (partial or complete) during the first 16 weeks on follow up as per investigator assessment of soft tissue/visceral disease per RECIST 1.1 in subjects who have a measurable tumour and/or Prostate Cancer Working Group 3 (PCWG3) criteria for bone metastases

SECONDARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | Through study completion, an average of 2 years
  Time from randomization to first objective evidence of radiographic progression, based on RECIST 1.1 for soft tissue/visceral disease and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines for bone metastases, or death, whichever occurs first.
Time to PSA Progression (TTPP) | Through study completion, an average of 2 years
  Time from randomization to PSA progression defined as PSA greater than or equal to 25 percent and greater than or equal to 2ng/mL from nadir (or baseline for participants with no PSA decline), confirmed by a second value obtained 3 or more weeks apart as per PCWG3 guidelines.
Time to unequivocal clinical progression (TTCP) | Through study completion, an average of 2 years
  Time from randomization to clinical worsening of prostate cancer related symptoms, as new onset cancer pain requiring chronic administration of opiate analgesia, deterioration from prostate cancer of Eastern Cooperative Oncology Group (ECOG) performance status score to 3 or higher, time to first skeletal-related event (the time from randomization to first incidence of radiotherapy to the bone or bone surgery, pathological bone fracture, spinal cord compression, or change of antineoplastic therapy to treat bone pain); or initiation of subsequent lines of active treatment including cytotoxic chemotherapy or radiation therapy or surgical intervention due to complications or symptoms related to disease progression.
Progression Free Survival (PFS) | Through study completion, an average of 2 years
  Time from randomization to PSA progression, unequivocal clinical progression or radiographic progression, whichever occurs first.
Incidence of adverse events (AEs) | Through study completion, an average of 2 years
  Total, grouped by grades and AEs category, related and unrelated with the trial treatment. The AEs Defined as incidence of prespecified AEs as per National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v.5.0, change from baseline in targeted vital signs and change from baseline in targeted clinical laboratory test results.
Incidence of serious adverse events (SAEs) | Through study completion, an average of 2 years
  Number of Serious Adverse Events, related and unrelated. SAEs leading to treatment discontinuation.
Drug compliance | Through study completion, an average of 2 years
  Percentage of dose taken for each treatment drug, dose reductions, dose discontinuation (temporary or permanent)

OTHER OUTCOMES:
Assessment of PSA response rate | Through study completion, an average of 2 years
  In participants with and without germline and/or somatic DDR alterations.
Assessment of ORR | Through study completion, an average of 2 years
  In participants with and without germline and/or somatic DDR alterations
Assessment of rPFS | Through study completion, an average of 2 years
  In participants with and without germline and/or somatic DDR alterations
Assessment of TTPP | Through study completion, an average of 2 years
  In participants with and without germline and/or somatic DDR alterations.
Assessment of TTCP | Through study completion, an average of 2 years
  In participants with and without germline and/or somatic DDR alterations.
Changes in expression levels of AR in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
Changes in expression levels of AR in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity
Changes in expression of AR-related genes in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
Changes in expression of AR-related genes in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity
Changes in open chromatin regions in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
Changes in open chromatin regions in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity
Survival signaling in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
Survival signaling in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity
DNA-damage in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
DNA-damage in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity
Deficient/proficient DNA-repair in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
Deficient/proficient DNA-repair in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity
Other biomarkers in tissue | Through study completion, an average of 2 years
  Changes from tissue samples, studying the correlation of these changes with clinical activity
Other biomarkers in plasma | Through study completion, an average of 2 years
  Changes from plasma samples, studying the correlation of these changes with clinical activity

CONTACTS AND LOCATIONS:
Overall Officials: Elena Castro, Dra., Principal Investigator — Hospital 12 de Octubre; Maria Ruiz Vico, Dra., Study Chair — Hospital 12 de Octubre; David Olmos, Dr., Study Chair — Hospital 12 de Octubre
Locations (12):
- Spain (12):
  - Institut Català d'Oncologia (ICO), Badalona, Barcelona
  - Consorcio Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Jerez de la Frontera, Cadiz, Cádiz
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario Del Mar., Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Miguel Servet, Zaragoza